CLINICAL TRIAL: NCT03782610
Title: Early Prediction of Spontaneous Patent Ductus Arteriosus (PDA) Closure and PDA-Associated Outcomes
Status: Active, not recruiting | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Ohio State University (Other); OhioHealth (Other); Mount Carmel Health System (Other)
Responsible Party: Principal Investigator, Jonathan Slaughter, Principal Investigator, Nationwide Children's Hospital
Other Study IDs: 1800684; 1R01HL145032 (NIH)
Record Dates: First submitted 2018-12-17; First posted 2018-12-20 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Patent Ductus Arteriosus; Preterm Infant; Bronchopulmonary Dysplasia; Neurodevelopmental Abnormality
Keywords: Patent Ductus Arteriosus; Preterm Infant; Echocardiogram; Prospective Cohort; Prediction Modeling
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth; Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 22 Months
Biospecimen Retention: Samples Without DNA — Serum biomarkers: beta-natriuretic peptide (BNP); N-terminal pro-B-type natriuretic peptide (NTpBNP)
  Urine biomarkers: neutrophil gelatinase-associated lipocalin (NGAL); heart-fatty acid-binding protein (H-FABP)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Study Cohort: 450 Infants
- Validation Cohort: 225 Infants. Will allow subsequent validation of models derived from the Primary Study Cohort.

SUMMARY:
Patent ductus arteriosus (PDA), very common in preterm infants, is the delayed closure of a fetal blood vessel that limits blood flow through the lungs. PDA is associated with mortality and harmful long term outcomes including chronic lung disease and neurodevelopmental delay. Although, treatments to close PDA likely benefit some infants, widespread routine treatment of all preterm infants with PDA may not improve important outcomes. Left untreated, most PDAs close spontaneously. Thus, PDA treatment is increasingly controversial and varies markedly between hospitals and individual providers. The relevant and still unanswered clinical question is not whether to treat all preterm infants with PDA, but whom to treat and when. Treatment detriments may outweigh benefits, since all forms of deliberate PDA closure have potential adverse effects, especially in infants destined for early, spontaneous PDA closure. Unfortunately, clinicians cannot currently predict in the 1st month which infants are at highest risk for persistent PDA, and which combination of clinical risk factors, echocardiographic (echo) measurements, and serum biomarkers may best predict PDA-associated harm. The American Academy of Pediatrics has acknowledged early identification of infants at high-risk from PDA as a key research goal for informing future PDA-treatment effectiveness trials.

Our objective is to use a prospective cohort of untreated infants with PDA to predict spontaneous ductal closure timing and identify echo measurements and biomarkers that are present in the 1st postnatal month and associated with long-term impairment. Our central hypothesis is that these risk factors can be determined to inform appropriate clinical treatments when necessary. Clinical, serum and urine biomarkers (BNP, NTpBNP, NGAL, H-FABP), and echo variables sequentially collected during each of the first 4 postnatal weeks will be examined. In addition myocardial deformation imaging (MDI) and tissue Doppler imaging (TDI), innovative echo methods, will facilitate the quantitative evaluation of myocardial performance. Aim 1 will estimate the probability of spontaneous PDA closure and predict the timing of ductal closure using echo, biomarker, and clinical predictors. Aim 2 will specify which echo predictors and biomarkers are associated with mortality and severity of respiratory illness at 36-weeks PMA. Aim 3 will identify which echo predictors and biomarkers are associated with 22- to 26-month neurodevelopment. All models will be validated in a separate cohort. This project will significantly contribute to clinical outcomes and PDA management by reducing unnecessary and harmful overtreatment of infants with a high probability of early spontaneous PDA closure, and will permit the development of outcomes-focused trials to examine the effectiveness of PDA closure in those "high-risk" infants most likely to receive benefit.

ELIGIBILITY:
Inclusion Criteria:

* Born between 23-weeks + 0 days (23_0/7 wks) and 29-weeks + 6 days (29_6/7 wks) gestation, inclusive
* Admitted to a study neonatal intensive care unit (NICU) within 72-hours of birth
* PDA noted on initial screening echo at <72 postnatal hours

Exclusion Criteria:

* Life-threatening congenital abnormalities, including congenital heart disease (other than PDA or small atrial septal defects/patent foramen ovale/muscular VSD)
* Parents have chosen to allow natural death (placed a do not resuscitate order)

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A cohort of consecutively enrolled preterm infants born between 23- and 30-weeks gestation with patent ductus arteriosus (PDA) documented on echocardiogram within 72-hours postnatal.
Sampling Method: Non-Probability Sample
Enrollment: 675 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Patent ductus arteriosus (PDA) closure documented via echocardiogram by 36-weeks postmenstrual age (PMA) (binary) | Outcome will be documented between <72-hour screening echo and 36-weeks PMA.
  Documented closure of PDA on echocardiogram. Echocardiograms to document the primary outcome will be conducted weekly for the first four postnatal weeks and every other week thereafter, between study entry and 36-weeks PMA until PDA-closure is documented
Mortality or supplemental oxygen or positive-pressure respiratory support at 36-weeks PMA (binary) | Outcome will be documented between <72-hour screening echo and 36-weeks PMA
  Death occurring between study entry at <72-hours postnatal and 36-weeks PMA OR an oxygen or positive-pressure ventilation requirement at 36-weeks gestational age (=moderate bronchopulmonary dysplasia [BPD] or severe BPD)
Composite Bayley III Motor Score at 22-26 months corrected age (continuous) | Bayley III Score Testing will occur at 22 to 26 months corrected age (CA) (age since birth - number of weeks born before 40-weeks gestation)
  Composite motor score at 22 to 26-months postnatal as measured by Bayley Scales of Infant and Toddler Development- 3rd Edition (Bayley III)

SECONDARY OUTCOMES:
Mortality by 36-weeks PMA (binary) | Death occuring between 72-hours postnatal and 36-weeks PMA
Bayley III Gross Motor Development Scaled Standard Score at 22-26 months corrected age (continuous) | Recorded at 22-26 months corrected age
Bayley III Fine Motor Development Scaled Standard Score postnatal age at 22-26 months corrected age (continuous) | Recorded at 22-26 months corrected age
Bayley III Cognitive Composite Score at 22-26 months corrected age (continuous) | Recorded at 22-26 months corrected age
Bayley III Language Composite Score at 22-26 months corrected age (continuous) | Recorded at 22-26 months corrected age

OTHER OUTCOMES:
Normal cardiac function at 36-weeks PMA (binary) | Recorded at 36-weeks PMA or discharge if prior to 36-weeks
  No functional abnormalities identified on the 36-week echocardiogram, as read by the study cardiologist
Quantitative myocardial deformation imaging (MDI) at 36-weeks PMA (continuous) | Recorded at 36-weeks PMA or discharge if prior to 36-weeks
Quantitative tissue Doppler imaging (TDI) at 36-weeks PMA (continuous) | Recorded at 36-weeks PMA or discharge if prior to 36-weeks
Pulmonary Hypertension at 36-weeks PMA (binary) | Recorded at 36-weeks PMA or discharge if prior to 36-weeks
  Pulmonary hypertension noted on the 36-week echocardiogram, as read by the study cardiologist
Normal left atrial size at 36-weeks PMA (binary) | Recorded at 36-weeks PMA or discharge if prior to 36-weeks
  No left atrial enlargement identified on the 36-week echocardiogram, as read by the study cardiologist
Normal left ventricular size at 36-weeks PMA (binary) | Recorded at 36-weeks PMA or discharge if prior to 36-weeks
  No left ventricular enlargement identified on the 36-week echocardiogram, as read by the study cardiologist
Normal right ventricular size at 36-weeks PMA (binary) | Recorded at 36-weeks PMA or discharge if prior to 36-weeks
  No right ventricular enlargement identified on the 36-week echocardiogram, as read by the study cardiologist
Oxygen Dependency (Moderate BPD) (binary) | Recorded at 36-weeks PMA
Positive-Pressure Dependency (Severe BPD) (binary) | Recorded at 36-weeks PMA
Length at 36-weeks PMA | Recorded at 36-weeks PMA or discharge if prior to 36-weeks
  Length in centimeters
General Movements Assessment (GMA) at 36-weeks corrected age | Recorded at 36-weeks PMA
  Prechtl's method for the qualitative assessment of general movements dysfunction
Time to enteral feed initiation | 72 hours postnatal to 36-weeks PMA
Time to a full enteral feed diet | 72 hours postnatal to 36-weeks PMA
  Infant is weaned from intravenous fluids to a full enteral feed diet (delivery of feeds may be via an enteric tube)
Oral feeding status (binary) | Recorded at 36-weeks PMA
  Infant is taking all feeds by mouth (PO feeds) by 36-weeks PMA
Weight at 36-weeks PMA | Recorded at 36-weeks PMA or discharge if prior to 36-weeks
  Weight in grams
Occipitofrontal circumference (OFC) at 36-weeks PMA | Recorded at 36-weeks PMA or discharge if prior to 36-weeks
  OFC in centimeters
Body Mass Index (BMI) at 36-weeks PMA | Recorded at 36-weeks PMA or discharge if prior to 36-weeks
  BMI calculated by (BMI= weight in kg/length in meters squared)
Supplemental oxygen or positive-pressure respiratory support at 40-weeks PMA (binary) | Recorded at 40-weeks PMA
Mortality by 22-26 months corrected age | Death occuring between 72-hours postnatal and 22-26 months corrected age
Duration of ductal patency from 72-hours postnatal until 22 to 26-months corrected age follow-up | 72 hours postnatal until 22-26 months follow-up visit
Supplemental oxygen support (binary) at 22-26 months corrected age | Recorded at 22-26 months study follow-up visit
Supplemental positive-pressure ventilation support (binary) at 22-26 months corrected age | Recorded at 22-26 months study follow-up visit
Weight at 22-26 months corrected age | Recorded at 22-26 months study follow-up visit
  Weight in kilograms
Length at 22-26 months corrected age | Recorded at 22-26 months study follow-up visit
  Length in centimeters
Body Mass Index (BMI) at 22-26 months corrected age | Recorded at 22-26 months study follow-up visit
  BMI calculated by (BMI= weight in kg/length in meters squared)
Feeding status via full oral feeding or gastric-tube (binary) at 22-26 months corrected age | Recorded at 22-26 months study follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan L Slaughter, MD, MPH, Principal Investigator — Nationwide Children's Hospital/The Ohio State University; Carl H Backes, MD, Principal Investigator — Nationwide Children's Hospital/The Ohio State University
Locations (4):
- United States (4):
  - Nationwide Children's Hospital Main Campus Neonatal Intensive Care Unit, Columbus, Ohio
  - Nationwide Children's Neonatal Intensive Care Unit at The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Nationwide Children's Neonatal Intensive Care Unit at OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - Nationwide Children's Hospital Neonatal Intensive Care Unit at OhioHealth Grant Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
We welcome the opportunity to share data from our investigation. All patient identifiers will be removed from the final dataset. Following the completion and publication of our investigation, we will make the data available to other users under a data sharing agreement. We will ask under the agreement that other users will commit to using the data only for research purposes, that they will not identify individual study subjects, that they will securely store the data electronically using password protection or encryption, that they will delete or destroy the data after the completion of their investigation, and that they will acknowledge the contribution of the funding agency (NIH NHLBI) and our investigative team in collecting the original data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available after the completion of our planned investigation and publication of the results. We anticipate the completion of the investigation and publication will occur by December 2025
Access Criteria: Email study co-PIs Jonathan Slaughter (Jonathan.Slaughter@nationwidechildrens.org) and Carl Backes (Carl.Backes@nationwidechildrens.org)

REFERENCES:
- [Background] Benitz WE; Committee on Fetus and Newborn, American Academy of Pediatrics. Patent Ductus Arteriosus in Preterm Infants. Pediatrics. 2016 Jan;137(1). doi: 10.1542/peds.2015-3730. Epub 2015 Dec 15. PMID 26672023
- [Background] Slaughter JL, Reagan PB, Newman TB, Klebanoff MA. Comparative Effectiveness of Nonsteroidal Anti-inflammatory Drug Treatment vs No Treatment for Patent Ductus Arteriosus in Preterm Infants. JAMA Pediatr. 2017 Mar 6;171(3):e164354. doi: 10.1001/jamapediatrics.2016.4354. Epub 2017 Mar 6. PMID 28046188
- [Background] Pavlek LR, Slaughter JL, Berman DP, Backes CH. Catheter-based closure of the patent ductus arteriosus in lower weight infants. Semin Perinatol. 2018 Jun;42(4):262-268. doi: 10.1053/j.semperi.2018.05.009. Epub 2018 Jun 13. PMID 29909074
- [Derived] Runte KE, Flyer JN, Edwards EM, Soll RF, Horbar JD, Yeager SB. Variation of Patent Ductus Arteriosus Treatment in Very Low Birth Weight Infants. Pediatrics. 2021 Nov;148(5):e2021052874. doi: 10.1542/peds.2021-052874. Epub 2021 Oct 21. PMID 34675131
- [Derived] Slaughter JL, Cua CL, Notestine JL, Rivera BK, Marzec L, Hade EM, Maitre NL, Klebanoff MA, Ilgenfritz M, Le VT, Lewandowski DJ, Backes CH. Early prediction of spontaneous Patent Ductus Arteriosus (PDA) closure and PDA-associated outcomes: a prospective cohort investigation. BMC Pediatr. 2019 Sep 13;19(1):333. doi: 10.1186/s12887-019-1708-z. PMID 31519154

DOCUMENTS (1):
  • Informed Consent Form (2018-12-26): https://cdn.clinicaltrials.gov/large-docs/10/NCT03782610/ICF_000.pdf